CLINICAL TRIAL: NCT05692752
Title: Expression of microRNA-133a and microRNA-208b in Acute Myocardial Infarction Egyptian Patients
Brief Title: Expression of microRNA-133a and microRNA-208b in Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Islamia University of Bahawalpur (Other)
Collaborators: German University in Cairo (Other)
Responsible Party: Principal Investigator, Hafiz Abdul Sattar Hashmi, Lecturer, Islamia University of Bahawalpur
Other Study IDs: UCCM/2022/EGT/01
Record Dates: First submitted 2022-12-22; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Myocardial Infarction, Acute
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test Group: The study group included 10 patients,
  1. men and women
  2. between age of 35-60 year
  3. chest pain lasting for at least 30 minutes,
  4. electrocardiogram (ECG) finding that display ST-segment elevation (STEMI)
  Interventions: Other: No intervention
- Control Group: The study group included 10 patients,
  1. men and women
  2. between age of 35-60 year
  3. having no complaint of health issue,
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Expression of miR-133a &208b at 4, 8, 12, 24 and 48 hours from the first appearance of myocardial infarction (MI) symptoms
  Other Names: Expression of miR-133a & 208b

SUMMARY:
Cardiac-enriched micro-RNAs (miRNAs), micro RNA 208b and 133a(MiR-208b, MiR-133a)) corresponds to the health and disorders of the cardiovascular system. An intron of the cardiac myosin heavy chain gene MYH7 encodes miR-208b. It is found on chromosome 14 in humans. Identify new diagnostic biomarkers based on miRNAs, researchers examine the expression of miR-133a and 208b at various time points (04 hours, 08 hours, 12 hours, 24 hours, 48 hours) following the development of the infarct and compared it to the traditional myocardial infarction biomarkers cardiac troponine (cTnl) and Creatine kinase-MB (CK-MB).

DETAILED DESCRIPTION:
The 98% of human genes are non-coding RNA, which is further divided into long non-coding RNA (lncRNA, > 200 bp) and short non-coding RNA (200 bp, including microRNA (miRNA) and circular RNA). More than 2000 human miRNAs have been discovered, and it seems that they regulate around 60% of human genes.Through a number of pathways, miRNAs control the development, re-modelling, and regeneration of the heart as well as endothelial function, vasculo-genesis, and neoangiogenesis. 30% of the genes in the human genome are regulated by about 1000 miRNAs. Endogenous miRNAs are 19-22 nucleotide single-stranded RNA molecules that frequently target the 3' untranslated regions (3'-UTR) of mRNAs to regulate gene expression at the post-transcriptional level in physiological processes, disease development, and conditions like cancer, autoimmune and inflammatory diseases, neuro-degenerative diseases, and cardiovascular diseases. Cardiac-enriched miRNAs, MiR-208 in health and disorders of the cardiovascular system are investigated.

Identify new diagnostic biomarkers based on miRNAs, researchers examine the expression of miR-133a and 208b at various time points (04 hours, 08 hours, 12 hours, 24 hours, 48 hours) following the development of the infarct and compared it to the traditional myocardial infarction biomarkers cTnl and CK-MB.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with ST-Elevated Myocardial Infarction will be identified at the Coronary Care Unit at Ain-shams University hospital
2. Acute episode of Myocardial Infarction
3. With No history of previous Myocardial Infarction Treatment

Exclusion Criteria:

1. Patients not diagnosed with ST-Elevated Myocardial Infarction and healthy at the Coronary Care Unit at Ain-shams 2. University hospital
2. Previously Known patients of Myocardial infacrtion
3. Previous medication

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient registering at the Coronary Care Unit at Ain-shams University hospital German University in Cairo, New Cairo City,.Egypt
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-14 (Actual)

PRIMARY OUTCOMES:
Expression of miR-133a | 04 hours from the onset of the infarct
  Expression during episodes of myocardial infarction
Expression of miR-133a | 08 hours from the onset of the infarct
  Expression during episodes of myocardial infarction
Expression of miR-133a | 12 hours from the onset of the infarct
  Expression during episodes of myocardial infarction
Expression of miR-133a | 24 hours from the onset of the infarct
  Expression during episodes of myocardial infarction
Expression of miR-133a | 48 hours from the onset of the infarct
  Expression during episodes of myocardial infarction
Expression of miR-208b | 04 hours from the onset of the infarct
  Expression during episodes of myocardial infarction
Expression of miR-208b | 08 hours from the onset of the infarct
  Expression during episodes of myocardial infarction
Expression of miR-208b | 12 hours from the onset of the infarct
  Expression during episodes of myocardial infarction
Expression of miR-208b | 24 hours from the onset of the infarct
  Expression during episodes of myocardial infarction
Expression of miR-208b | 48 hours from the onset of the infarct
  Expression during episodes of myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Sally I Hassanien, Ph.D, Principal Investigator — Biochemistry Department German University in Cairo, 11835, Cairo, Egypt; Hafiz A Sattar, M.Phil, Principal Investigator — University College of Conventional Medicine, The Islamia University of Bahawalpur, Punjab, Pakistan
Locations (1):
- Biochemistry Department, Faculty of Pharmacy and Biotechnology, German University in Cairo, Main Entrance Al Tagamoa Al Khames, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
De-identified data will be published.